CLINICAL TRIAL: NCT01347918
Title: Small Intestinal Transit and Motor Function in Health and IBS Patients Studied by Combined 1H and 19F Magnetic Resonance Imaging
Brief Title: 1H-19F Gastrointestinal MRI in Health and IBS
Status: Suspended | Type: Observational
Why Stopped: Technical problems
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: GI-MRI; 2011-MD-0005 (Other: Swissmedic)
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Fluorine MRI, small intestinal transit and motor activity
MeSH Terms: conditions — Irritable Bowel Syndrome; Motor Activity | interventions — Karaya Gum; Normacol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: Healthy controls
  Interventions: Device: 19F capsule; Dietary Supplement: sterculia
- IBS: Patients that fulfil the Rome III criteria for irritable bowel syndrome (IBS)
  Interventions: Device: 19F capsule; Dietary Supplement: sterculia

INTERVENTIONS:
Device: 19F capsule — Two 19F capsules, one filled with hexafluorobenzene (HFB) and the other filled with perfluoro-15-crown-5-ether (PCE) will be administered orally together with 100 ml of water.
  Other Names: fluorine labeled capsule
Dietary Supplement: sterculia — 7g of sterculia will be ingested over one week together with the normal breakfast.
  Other Names: Normacol

SUMMARY:
The aim of this project is to demonstrate and validate the ionizing radiation free and non invasive assessment of small intestinal anatomy, content and function in healthy and disease by a newly developed combined proton (1H) and fluorine (19F) magnetic resonance imaging (MRI) framework. Meal induced and pathology related alterations in small intestinal motor activity, gas distribution and anatomy of healthy volunteers and patients with irritable bowel syndrome (IBS) will be analyzed with this non invasive MRI approach.

The multinuclear imaging framework consists of a 1H and 19F capable clinical 3T MRI system with standard 1H abdominal surface coils, a dual-channel transmit-receive abdominal 19F surface coil, fluorine labelled impermeable and biocompatible capsules for oral administration (19F capsule) and a 19F projection imaging sequence allowing for the non-invasive detection of the gastrointestinal positions of single and multiple ingested capsules in real time. Dedicated post-processing algorithms are applied to extract parameters of intestinal motor activity from the detected intraluminal capsule movements.

The proposed unique imaging modality allows for the concurrent, non invasive and repeated analysis of important physiologic parameters of intestinal function together with detailed anatomical information and thus presents an ideal tool for the evaluation of the analyzed parameters as potential biomarkers in IBS.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* Healthy volunteers and IBS patients must fill out the validated Birmingham IBS Symptom Questionnaire
* Healthy volunteers must be symptom free of any abdominal complaints.
* IBS patients are defined based on clinical symptoms as described in the Rome III criteria for irritable bowel syndrome:

  * Symptoms of recurrent abdominal pain or discomfort and a marked change in bowel habit for at least six months, with symptoms experienced on at least three days of at least three months. Two or more of the following must apply:
* Pain is relieved by bowel movement
* Onset of pain is related to a change in frequency of stool
* Onset of pain is related to a change in the appearance of stool
* Written informed consent

Exclusion criteria:

* Age under 18 or above 65
* Pathologic underweight or overweight (BMI <18 or >30kg/m2)
* Previous history of gastrointestinal disease or surgery (excludes appendectomy, cholecystectomy, hernia repair and anorectal disorders)
* Previous cardiorespiratory (excludes arterial hypertension), hematologic, renal, atopic, alimentary or psychiatric disease, diabetes, drug or alcohol abuse, psychiatric disease
* Patient unable to stop medication that alters gut function for 72 hours prior to the study, including anticholinergics, prokinetics, proton-pump inhibitors, non-steroidal antiinflammatory drugs
* Presence of metallic implants, devices or metallic foreign bodies
* Pregnancy and lactation (female patients of child bearing age will receive a pregnancy test prior to study)
* Female volunteers without adequate contraception for the duration of the study Involvement in any other clinical trial during the course of this trial, nor within a period of 30 days prior to its beginning or 30 days after its completion
* Allergy against silicone
* Claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The healthy controls will be selected from among students and volunteers that have responded to advertisments in local notice boards of the Zurich University Hospital and the University of Zurich, as well as in an email newsletter ("Mediflash") of the Medical Student Organisation.
  The IBS patients are selected from the patient population seen in the Klinik and Polyklink für Innere Medizin at the University Hopsital Zurich.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Small intestinal transit time in minutes | Regularly over 4 hours

SECONDARY OUTCOMES:
Small intestinal length and intestinal course | at 4 hours
Small intestinal motor activity index | At 4 hours
Small intestinal transport velocity | Regularly over 4 hours
Local intestinal residence times | Regularly over 4 hours.
Volume and distribution of intestinal gas | Regularly over 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Schwizer, Prof. MD, Principal Investigator — University Hospital Zurich, Gastroenterology & Hepatology
Locations (1):
- University Hospital Zurich, Gastroenterology, Zurich, Switzerland